CLINICAL TRIAL: NCT04169698
Title: Evaluation of the Efficacy and Tolerability of Alendronate Versus Denosumab in Kidney Transplant Patients With Reduced Bone Mineral Density
Brief Title: Alendronate Versus Denosumab in Kidney Transplant Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Collaborators: Nahda University (Other)
Responsible Party: Principal Investigator, Sherihan Ahmed Sayed Omar, Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHCL236
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis, Osteopenia; Renal Transplant Recipient
Keywords: Denosumab; Alendronate; Osteoporosis; renal transplant
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Denosumab; Alendronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (No Intervention): Participants will receive daily supplements of calcium (1000 mg), vitamin D (800 IU or more) and calcitriol (0.25 micro gram).
- Denosumab group (Experimental): Participants will receive a single 60 mg subcutaneous dose of denosumab (Prolia) every 6 months for 12 months plus daily supplements of calcium (1000 mg), vitamin D (800 IU or more) and calcitriol (0.25 micro gram).
  Interventions: Drug: Denosumab 60 mg/ml [Prolia]
- Alendronate group (Experimental): Participants will receive an oral alendronate at a dose of 70 mg once every week for up to 12 months plus daily supplements of calcium (1000 mg), vitamin D (800 IU or more) and calcitriol (0.25 micro gram).
  Interventions: Drug: Alendronate 70Mg Tab

INTERVENTIONS:
Drug: Denosumab 60 mg/ml [Prolia] — full length human monoclonal antibody against the receptor activator of nuclear factor kappa-B ligand
  Arms: Denosumab group
Drug: Alendronate 70Mg Tab — Bisphosphonates
  Arms: Alendronate group

SUMMARY:
The management of bone disease has often been neglected post-transplantation, when the clinical focus is on allograft function and immunological sequelae. However, most renal transplant recipients (RTRs) have pre-existing CKD-MBD, which results in changes to mineral metabolism and reduced bone mineral density (BMD) and quality, which are linked to an increased incidence of fractures and cardiovascular disease. Bone loss is greatest in the first 6-12 months post-transplantation, during which period any intervention is likely to be of greatest benefit. Anti-resorptive agents all inhibit bone resorption. Since bisphosphonates and densoumab are the most widely used anti-resorptive agents for osteoporosis, we conduct this prospective interventional comparative study to compare the efficacy and tolerability of alendronate versus denosumab in de novo kidney transplant recipients with reduced bone mineral density, in the first 12 months treatment after kidney transplantation.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) exhibit a complex form of bone disease defined by KDIGO as "Mineral and Bone Disorder" (CKD-MBD). CKD-MBD generally encompasses two pathological disorders, namely vascular calcification and renal osteodystrophy, which is the bone health impairment associated with chronic kidney disease. Among the complications associated with renal osteodystrophy, hip or vertebral fractures are associated with an increase in morbidity and mortality in patients with end-stage kidney disease.

CKD-MBD is a systemic disease that links disorders of mineral and bone metabolism due to CKD to either one or all of the following: abnormalities of calcium, phosphorus, parathyroid hormone or vitamin D metabolism; abnormalities in bone turnover, mineralization, volume, linear growth or strength; or vascular or other soft-tissue calcification. Consequently, since bone status in recently transplanted patients reflects several years of CKD-MBD, it would be useful to assess bone status in this population.

The management of bone disease has often been neglected post-transplantation, when the clinical focus is on allograft function and immunological sequelae. However, most renal transplant recipients (RTRs) have pre-existing CKD-MBD, which results in changes to mineral metabolism and reduced bone mineral density (BMD) and quality, which are linked to an increased incidence of fractures and cardiovascular disease. Pre-existing renal osteodystrophy, including adynamic bone disease, is further affected post-transplantation by the use of immunosuppressive medications (glucocorticoids and calcineurin-inhibitors), variable renal allograft function and post-transplantation diabetes mellitus.

Successful renal transplantation corrects many metabolic abnormalities associated with the development of renal osteodystrophy. However, osteopenia and osteoporosis remain prevalent, even in patients with well-functioning grafts. Increasing attention has focused on preventing late complications of transplantation and on patient quality of life by addressing factors affecting long-term morbidity, such as cardiovascular risk, post-transplantation diabetes mellitus, cancer, and bone disease.

The spectrum of bone diseases in kidney transplant recipients includes renal osteodystrophy, osteoporosis, bone fracture, and osteonecrosis. Earlier studies after transplantation indicate that BMD declines by 4%-10% in the first 6 months, with a further decrease of 0.4%-4.5% in lumbar BMD between 6 and 12 months. After 1 year, BMD remains relatively stable with no further decline but at significantly lower levels than healthy controls. This reduction in BMD contributes to an increased risk of fractures.

Osteoporosis is defined as skeletal disorder characterized by compromised bone strength with low BMD and bone quality predisposing to an increased risk of fracture and bone fragility. Osteoporosis has also been defined quantitatively using BMD and can be expressed as standard deviation (SD) score comparing an individual's BMD with that of a reference population as measured by dual x-ray absorptiometry (DEXA). A T-score that is ≤ -2.5 is indicative of osteoporosis.

In RTRs, a noninvasive cost-effective tool regarding diagnostic evaluation of osteoporosis is BMD monitoring with DEXA scans. BMD is the amount of bone mass per unit volume (volumetric density), or per unit area (areal density), and both can be measured in vivo by densitometric techniques. A wide variety of techniques is available to assess bone mineral that are reviewed elsewhere. The most widely used are based on X-ray absorptiometry of bone, particularly dual energy X-ray absorptiometry, since the absorption of X-rays is very sensitive to the calcium content of the tissue of which bone is the most important source.

DEXA is obtained by aiming two radiograph beams with different energy levels at the patient's bones. After subtracting the soft tissue absorption, the BMD is determined. DEXA is the most widely used noninvasive technique for measuring BMD in the general population. Low BMD by DEXA is a robust and consistent risk factor for fracture and treatments that increase BMD reduce fracture risk.

Bone mineral density is most often described as a T- or Z score, both of which are units of SD. The T-score describes the number of SDs by which the BMD in an individual differs from the mean value expected in young healthy individuals. The Z-score describes the number of SDs by which the BMD in an individual differs from the mean value expected for age and sex. It is mostly used in children and adolescents.

Bone loss is greatest in the first 6-12 months post-transplantation, during which period any intervention is likely to be of greatest benefit. Anti-resorptive agents all inhibit bone resorption. The FDA-approved anti-resorptive agents include calcitonin, estrogens, selective estrogen receptor modulators, bisphosphonates and denosumab. Each anti-resorptive agent has each owns unique mechanism of action. Since bisphosphonates and densoumab are the most widely used anti-resorptive agents for osteoporosis, these two agents will be focused here.

There is strong evidence that bisphosphonates prevent post-transplantation bone loss; however, data are lacking that this clearly extends to a reduction in fracture incidence. Denosumab is a potential alternative to vitamin D receptor agonists and bisphosphonates in reducing post-transplantation bone loss; however, further studies are needed to demonstrate its safety in patients with a significantly reduced estimated glomerular filtration rate (eGFR). Clinical judgement remains the cornerstone of this complex clinical problem, providing a strong rationale for the formation of combined endocrinology and nephrology clinics to treat patients with Chronic Kidney Disease-Mineral and Bone Disorder, before and after transplantation.

Bisphosphonates are chemical analogues of naturally occurring pyrophosphates (P-O-P), degradation products of adenosine triphosphate metabolism. Pyrophosphates are rapidly metabolized by the ubiquitous presence of pyrophosphatases, while bisphosphonates (P-C-P) are not metabolized. Once entering the blood stream, bisphosphonates are rapidly taken up by bone, the only tissue that binds bisphosphonates. In bone, bisphosphonates inhibit bone resorption by two mechanisms: a physiochemical one stabilizing the calcium-phosphorus surface and a cellular one by inhibiting osteoclast activity. Bisphosphonates are cleared by the kidney both by filtration and active proximal tubular secretion. Bisphosphonates are retained in bone in the remodeling resorption cavity and the amount of bisphosphonate retained in probably a function of the baseline remodeling space, the chronic rate of bone turnover and the glomerular filteration rate (GFR). While oral bisphosphonates are poorly (less than 1% of a single dose) absorbed and 50% of that excreted unchanged by the kidney, intravenous bisphosphonate show a 100% bioavailability with still 50% of an intravenous dose excreted by the kidney. Treatment with bisphosphonates before and after renal transplantation had a favorable effect on BMD, with bisphosphonates, such as pamidronate and alendronate, being preferable to other treatments.

Denosumab is a full length human monoclonal antibody against the receptor activator of nuclear factor kappa-B ligand (RANKL), a cytokine that is essential for the formation, function, and survival of osteoclasts. By binding RANKL, denosumab prevents the interaction of RANKL with RANK on osteoclasts and reversibly inhibits osteoclast-mediated bone resorption. It was approved by the U.S. Food and Drug Administration in June 2010 as a new treatment for postmenopausal osteoporosis in women who are at high risk of fractures. Denosumab is not renally cleared, which makes it more attractive than bisphosphonates in patients with significant graft dysfunction, although there are little data of its use in the transplant population. Denosumab treatment may be useful to improve bone health in the first year after kidney transplantation and was safe except for a higher number of urinary tract infections and asymptomatic episodes of hypocalcemia.

There are no comparative studies of different agents available for treatment of RTRs, who remain a heterogeneous population in terms of renal function. However, given that bone loss is greatest in the first 12 months, any benefit will be greatest in this period. KDIGO 2017 guidelines suggest treatment with vitamin D, calcitriol/alfacalcidol, and/or antiresorptive agents be considered in patients in the first 12 months after kidney transplant with an estimated glomerular filtration rate greater than approximately 30 ml/min/1.73 m2 and low BMD.

Finally, this prospective interventional comparative study will be conducted to compare the efficacy and tolerability of alendronate versus denosumab in de novo kidney transplant recipients with reduced bone mineral density, in the first 12 months treatment after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 year old and medically stable.
* Recent kidney transplantation (up to 3 months).
* Stabilization of renal allograft function.
* Normal liver function.
* Reduced bone mineral density at least one SD lower than normal level for the same age and gender (T-score < -1).

Exclusion Criteria:

* Poor or unstable graft function (creatinine >200 lmol/L).
* Skeletal malignancies or bone metastases.
* Risk for osteosarcoma, such as Paget's disease of the bone.
* Unstable medical condition.
* Pregnancy and lactation.
* Autoimmune diseases.
* Predisposition to drug hypersensitivity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Bone mineral density measured by DEXA scan | One year
  Subject percent changes of bone mineral density at the lumbar spine, proximal femur and distal one-third radius from baseline to 6 and 12 months.

SECONDARY OUTCOMES:
Fracture incidence | One year
  The number of new clinical vertebral or non-vertebral fractures that are reported at any post baseline visit and subsequently confirmed by radiographs.
Graft function | One year
  Calculating the estimated GFR with the creatinine-based Chronic Kidney Disease Epidemiology Collaboration formula.
serum parathyroid hormone and vitamin D | One year
  parathyroid hormone and vitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Sherihan A Omar, Principal Investigator — Ain Shams University
Locations (1):
- National institute of urology and nephrology, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sayed SA, El Wakeel LM, Elseasi AM, Shawki MA. Evaluation of the efficacy and tolerability of alendronate versus denosumab in kidney transplant patients with reduced bone mineral density. Pharmacotherapy. 2023 Sep;43(9):904-912. doi: 10.1002/phar.2838. Epub 2023 Jun 22. PMID 37323099